CLINICAL TRIAL: NCT00763490
Title: Trial Of Double Umbilical Cord Blood Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: umcc 2007.137; HUM00017515 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-11

CONDITIONS: Hematological Malignancies
Keywords: umbilical cord blood; stem cell transplant; leukemia; multiple myeloma; lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Multiple Myeloma; Lymphoma | interventions — Stem Cell Transplantation; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Double cord blood transplant (Experimental): 'full intensity, double umbilical cord, stem cell transplant' with 'Flu/Bu4 conditioning regimen'
  Interventions: Procedure: Full intensity, double umbilical cord, stem cell transplant; Drug: Flu/Bu4 conditioning regimen; Radiation: Total Lymphoid Irradiation (TLI); Drug: Graft versus Host Disease prevention (GVHD prophylaxis); Drug: Mycophenolate Mofetil

INTERVENTIONS:
Procedure: Full intensity, double umbilical cord, stem cell transplant — stem cell transplant using two umbilical cord blood units, combined with a Flu/Bu4 conditioning regimen prior to transplantation
Drug: Flu/Bu4 conditioning regimen — Fludarabine: 40 mg/m² daily on days -5, -4, -3, -2
  Busulfan: 3.2 mg/kg IV daily on days -5, -4, -3, -2
Radiation: Total Lymphoid Irradiation (TLI) — one dose, 400 cGy,on day -1 or day 0, prior to cord blood infusion
Drug: Graft versus Host Disease prevention (GVHD prophylaxis) — Tacrolimus for GVHD (Graft Versus Host Disease Prevention) Tacrolimus - will begin on day -3 (IV or oral) for at least 180 days. Target trough level for tacrolimus is 8-12 ng/ml. In the absence of GVHD, tacrolimus tapering will begin on day +56 post transplant.
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil (MMF) for GVHD prophylaxis. MMF - will be given at a dose of 10mg/kg IV q 8 hours if the patient weight is more than 50 kg, or 15 mg/kg IV q 8 hours if less than 50 kg, beginning the morning of day -3. (If renal failure and Glomerular Filtration Rate (GFR) < 25 mL/min, the dose should not exceed 1 gm every 8 hours. (No dose adjustment for liver disease is required.) MMF should be given via IV until oral medications are tolerated.
  MMF will be stopped at Day +28 if no acute GVHD is seen by that time. If there is not any donor cell engraftment, MMF will be continued as directed by the attending physician. If the patient has active acute GVHD requiring systemic therapy, MMF may be continued.

SUMMARY:
This pilot research study is to investigate the safety and effectiveness of stem cell transplantation to treat blood-related (hematopoietic) cancers, using stem cells collected from two different, umbilical cord blood donors. Subjects in this study are receiving a stem cell transplant because other treatments have failed or their disease is unlikely to respond to other treatment options.

Blood-related cancers can be treated and sometimes cured with very high doses of chemotherapy and radiation therapy, given to kill the cancer cells; however, these treatments can prove unsuccessful and can harm normal cells in the bone marrow or a patient's disease may be unlikely to respond to these treatment options.

Hematopoietic stem cells transplantation (HSCT) is a potential cure, but opportunities to perform HSCT are limited by donor availability. Only 20-30% of patients may have matched family donors. In some cases, a mismatched family donor may be suitable. For patients needing a transplant who do not have a suitably matched family donor, blood stem cells from matched unrelated donors can be used. The length of time required to identify a matched unrelated donor presents another obstacle for patients waiting to receive an HSCT.

Blood stem cells are found in umbilical cord blood (UCB), which is blood left over in the placenta (afterbirth) after a baby is born. Usually this blood is discarded with the placenta, but over the past 15 years, we have learned how to collect and freeze cord blood cells to be used for transplants at a later time. A cord blood unit is the cord blood cells collected and stored from a single placenta. More than 6,500 umbilical cord blood stem cell transplants have been done worldwide, mostly in children with leukemia. One important factor affecting the success of a cord blood transplant is the cell dose (number of stem cells in the cord blood unit / recipient's weight). Patients who receive a high cell dose (> 2.5 x 107 cells/kilogram) have better marrow recovery and a higher rate of survival than those who receive a lower cell dose.

In an attempt to make UCB transplantation possible for bigger children, adolescents and adults, researchers have tried giving two cord blood units on the same day for their transplant, one after the other. The data from more than 150 "double cord blood" transplants in adults suggest that the "double cord blood" transplants may allow bone marrow recovery and survival in patients who do not have a single cord blood unit with enough cells for successful transplantation.

This is a pilot study to research the safety and effectiveness of using two UCB units in adult and pediatric UCB transplantation when combined with a conditioning regimen called Flu/Bu4/TLI (consisting of fludarabine, busulfan and total lymphoid irradiation).

ELIGIBILITY:
Inclusion Criteria:

* The candidate must have an incurable hematological malignancy or non-malignant hematological disorder and be eligible for transplant by the University of Michigan program.
* The candidate must have a life expectancy of less than one year without transplantation.
* The candidate must have two partially HLA-matched UCB (cord blood) units.Units must be HLA-matched minimally at 4 of 6 HLA-A and B (at intermediate resolution by molecular typing) and DRB1 (at high resolution by molecular typing) loci. Units must be HLA-matched at 3 of 6 HLA- A, B, DRB1 loci with each other (using same resolution of molecular typing as indicated above).
* The candidate must have access to two appropriately HLA-matched units that are available such that one unit delivers a pre-cryopreserved nucleated cell dose of at least 2.5 x 107 per kilogram and the second unit at least 2.0 x 107 per kilogram.

Exclusion Criteria:

* The candidate is an adult or pediatric patient who has a suitable related or unrelated donor available for transplant. Suitable donors include 8/8 (HLA-A,B,C and DR, with all loci high-resolution typing) or 7/8 related or unrelated donor available within 42 days of search initiation.
* The candidate has a Karnofsky (Adult) or Lansky (Pediatrics) performance status of < 70% at the time of admission for HSCT.
* The candidate is a patient with evidence of HIV infection.
* The candidate is a patient with active bacterial, fungal or viral infection not responding to treatment. Non-response to treatment is determined by body temperature, blood culture results, and radiographic findings as applicable.
* The candidate is pregnant.
* The candidate has any medical comorbidities/conditions that, in the opinion of the transplant team, would keep the patient from complying with the needs of the protocol and/or would markedly increase the morbidity and mortality from the procedure.
* The candidate has any conditions, in the opinion of the transplant team, such as substance abuse, or severe personality disorder that would keep the patient from complying with the needs of the protocol and would markedly increase the morbidity and mortality from the procedure.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Couriel, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Abedin S, Peres E, Levine JE, Choi S, Yanik G, Couriel DR. Double umbilical cord blood transplantation after novel myeloablative conditioning using a regimen of fludarabine, busulfan, and total lymphoid irradiation. Biol Blood Marrow Transplant. 2014 Dec;20(12):2062-6. doi: 10.1016/j.bbmt.2014.07.014. Epub 2014 Jul 18. PMID 25046834

RESULTS

PARTICIPANT FLOW:
Groups:
- Double Cord Blood Tranplant: Full intensity, double umbilical cord, stem cell transplant: stem cell transplant using two umbilical cord blood units, combined with a Flu/Bu4 conditioning regimen prior to transplantation.
Period: Overall Study
Arm/Group | Double Cord Blood Tranplant
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Double Cord Blood Tranplant
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 41 [11 to 64]
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive at 1 Year After Transplant
Description: One-year survival rate after transplant
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double Cord Blood Tranplant
Number analyzed (Participants) | 20
percentage of participants | 40 [19 to 60]

2. Secondary Outcome: Percentage of Patients Alive at the End of the Trial
Description: Event Free Survival (EFS) was determined. Patients were followed up to 5 years (median time of 2.35 years).
Time Frame: 5 Years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Double Cord Blood Tranplant
Number analyzed (Participants) | 20
percentage of patients | 35 [16 to 55]

3. Secondary Outcome: Cumulative Incidence of Neutrophil and Platelet Engraftment
Description: The failure to achieve a neutrophil count > 500/uL or a platelet count >30.0 x 10e9 /L within 35 days of the stem cell infusion will be defined as primary engraftment failure.
Time Frame: Day 35
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double Cord Blood Tranplant
Number analyzed (Participants) | 20
percentage of participants
  Cumulative incidence of platlet engraftment | 73 [48 to 88]
  Cumulative incidence of neutrophil engraftment | 89 [64 to 97]

4. Secondary Outcome: Incidence of Acute (Grade II-IV) and Chronic Graft-vs-host Disease(GVHD)
Description: The percentage of patients with acute GVHD (Grade II-IV) was determined at 100 days. Patients were followed up to 5 years and the percentage of patients that developed chronic GVHD at the end of the study was tabulated.
  Acute GVHD is staged and graded (grade 0-IV, where grade 0 is no involvement and involvement increases by grade) by the number and extent of organ involvement. Patients can have involvement of three organs: skin (rash/dermatitis), liver (hepatitis/jaundice), and gastrointestinal tract (abdominal pain/diarrhea).
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Double Cord Blood Tranplant
Number analyzed (Participants) | 20
percentage of patients
  Acute GVHD (Grades II-IV) | 40 [19 to 60]
  Chronic GVHD | 35 [16 to 65]

ADVERSE EVENTS:
Arm/Group | Double Cord Blood Tranplant
Serious Adverse Events (participants affected / at risk) | 14/20
Other Adverse Events (participants affected / at risk) | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Cord Blood Tranplant (N=20)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 3 (3)
Hypotension (Cardiac disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (3)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (2)
Infection with normal ANC (Infections and infestations) | 2 (2)
Confusion (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder spasms (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 2 (2)
Syndromes - Other (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Cord Blood Tranplant (N=20)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 3 (3)
Hypertension (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 6 (6)
Weight gain (Investigations) | 2 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection with normal ANC (Infections and infestations) | 3 (3)
Confusion (Nervous system disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Head Pain (Nervous system disorders) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cystitis (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No